CLINICAL TRIAL: NCT00971711
Title: Phase I, Open Label Safety Study of VSL#3 in Adults With Irritable Bowel Syndrome
Brief Title: Safety Study of Probiotics in Adults With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Robert Shulman, M.D., Professor of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24041; R01NR005337 (NIH); 005337
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; irritable bowel syndrome; abdominal pain; urgency; bloating; diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Diarrhea | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotic (Experimental): To determine the safety and effectiveness of the probiotic VSL#3 in adults with irritable bowel syndrome (IBS).
  Interventions: Biological: Probiotic

INTERVENTIONS:
Biological: Probiotic — The subjects will be randomized into either a 4 week or 8 week treatment period with the probiotic. The treatment will be open label. They will take 2 packets once daily.
  Other Names: VSL#3

SUMMARY:
Determine the safety and preliminary effectiveness of VSL#3 in adults with IBS.

DETAILED DESCRIPTION:
Recent studies performed outside the U.S. and/or prior to recent FDA requirements suggest that the probiotics in VSL#3 may be effective in IBS in adults. Because there is a significant unmet need for improved IBS therapies to prevent frequent exacerbations that lead to unscheduled health care, we will conduct a safety study of the probiotic VSL#3. Preliminary studies suggest that probiotics such as VSL#3 are effective in the treatment of adults with IBS but safety studies have not been carried out. A safety study of VSL#3 has been carried out in adult asthmatics that demonstrated no significant adverse effects. Before a trial of VSL#3 can be performed in children with IBS, the FDA has requested that a safety trial be conducted in adults with IBS.

Consent will be obtained from the subject.

Adults who meet the criteria for irritable bowel syndrome will be recruited and studied. They will have been diagnosed by an adult gastroenterologist.

During a baseline one week period, the subjects will keep a diary of pain episodes, pain severity, pain-induced interference with activity, and stooling pattern (i.e., pain/activity/stool diary).

Following the baseline period, the subjects will be randomized into either a 4 week or 8 week treatment period with the probiotic. The treatment will be open label. During the treatment period, subjects will keep the diary for pain and stooling habits and a daily record of symptoms (i.e., daily temperature monitoring).

At the end of the treatment period the pain/stool/activity diary will be repeated. Four weeks after the treatment period ends a follow-up phone call will be made to participants to check on their pain and stooling patterns.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise well and meet the criteria for IBS as defined by the Rome III criteria
* Ability to speak and understand English
* Telephone access
* IBS Severity Scale score of >= 75

Exclusion Criteria:

* Organic disease accounting for GI symptoms.
* Chronic illness such as renal disease, congenital heart disease, diabetes, moderate or severe asthma, abdominal surgery, or immunosuppressed (e.g., organ transplant recipient).
* Have received extraneous probiotic (i.e., not in a food such as yogurt) within 4 months of starting the study.
* Subjects who are taking prescription or over-the-counter medications for GI disorders that completely relieve their symptoms because by definition these individuals do not have IBS (e.g., antacids, proton pump inhibitors, histamine receptor antagonists).
* Medication allergies or contraindications which would preclude antimicrobial treatment for potential infection with VSL#3 component organisms.
* Pregnancy.
* Subjects who have an individual in the household who is immunosuppressed (e.g., genetic immune disorder, organ transplant).
* Oral temperature > 38.0 degrees Celsius.
* Poorly controlled hypertension, history of cardiac disease, stroke/cerebral vascular accident, bowel ischemia, or other risk factors for bowel ischemia.
* History of acute or chronic pancreatitis
* Cardiac valvular disease or other risk factor for endocarditis
* Subjects who indicate on the IBS scoring questionnaire that their pain is "severe" or "very severe."
* Subjects who pain lasts more than 5 out of 10 days.
* Subjects whose scores indicate more than mild IBS who are over 45 years of age

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety | Daily for 4 or 8 weeks of treatment and 1 month after treatment

SECONDARY OUTCOMES:
Pain and Stooling Improvement | 4 or 8 weeks of treatment and 1 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shulman, M.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor Clinic, Houston, Texas
  - Univerisity of Washington, Seattle, Washington

REFERENCES:
- [Background] Shulman RJ, Eakin MN, Jarrett M, Czyzewski DI, Zeltzer LK. Characteristics of pain and stooling in children with recurrent abdominal pain. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):203-8. doi: 10.1097/01.mpg.0000243437.39710.c0. PMID 17255832
- [Background] Thakkar K, Gilger MA, Shulman RJ, El Serag HB. EGD in children with abdominal pain: a systematic review. Am J Gastroenterol. 2007 Mar;102(3):654-61. doi: 10.1111/j.1572-0241.2007.01051.x. PMID 17222318
- [Background] Czyzewski DI, Eakin MN, Lane MM, Jarrett M, Shulman RJ, M D. Recurrent Abdominal Pain in Primary and Tertiary Care: Differences and Similarities. Child Health Care. 2007 May 2;36(2):137-153. doi: 10.1080/02739610701334970. No abstract available. PMID 20357915
- [Background] Lane MM, Weidler EM, Czyzewski DI, Shulman RJ. Pain symptoms and stooling patterns do not drive diagnostic costs for children with functional abdominal pain and irritable bowel syndrome in primary or tertiary care. Pediatrics. 2009 Mar;123(3):758-64. doi: 10.1542/peds.2008-0227. PMID 19254999
- [Background] Jarrett M, Heitkemper M, Czyzewski DI, Shulman R. Recurrent abdominal pain in children: forerunner to adult irritable bowel syndrome? J Spec Pediatr Nurs. 2003 Jul-Sep;8(3):81-9. doi: 10.1111/j.1088-145x.2003.00081.x. PMID 12942886
- [Background] Burr RL, Motzer SA, Chen W, Cowan MJ, Shulman RJ, Heitkemper MM. Heart rate variability and 24-hour minimum heart rate. Biol Res Nurs. 2006 Apr;7(4):256-67. doi: 10.1177/1099800405285268. PMID 16581896
- [Background] McOmber ME, Shulman RJ. Recurrent abdominal pain and irritable bowel syndrome in children. Curr Opin Pediatr. 2007 Oct;19(5):581-5. doi: 10.1097/MOP.0b013e3282bf6ddc. PMID 17885479
- [Background] Kellermayer R, Tatevian N, Klish W, Shulman RJ. Steroid responsive eosinophilic gastric outlet obstruction in a child. World J Gastroenterol. 2008 Apr 14;14(14):2270-1. doi: 10.3748/wjg.14.2270. PMID 18407608
- [Background] McOmber MA, Shulman RJ. Pediatric functional gastrointestinal disorders. Nutr Clin Pract. 2008 Jun-Jul;23(3):268-74. doi: 10.1177/0884533608318671. PMID 18595859
- [Background] Shulman RJ, Eakin MN, Czyzewski DI, Jarrett M, Ou CN. Increased gastrointestinal permeability and gut inflammation in children with functional abdominal pain and irritable bowel syndrome. J Pediatr. 2008 Nov;153(5):646-50. doi: 10.1016/j.jpeds.2008.04.062. Epub 2008 Jun 9. PMID 18538790
- [Derived] Boonma P, Shapiro JM, Hollister EB, Badu S, Wu Q, Weidler EM, Abraham BP, Devaraj S, Luna RA, Versalovic J, Heitkemper MM, Savidge TC, Shulman RJ. Probiotic VSL#3 Treatment Reduces Colonic Permeability and Abdominal Pain Symptoms in Patients With Irritable Bowel Syndrome. Front Pain Res (Lausanne). 2021 Sep 22;2:691689. doi: 10.3389/fpain.2021.691689. eCollection 2021. PMID 35295488
- See also: Clinical Trial For Children with Irritable Bowel Syndrome — http://clinicaltrials.gov/ct2/show/NCT00526903?term=NCT00526903&rank=1